CLINICAL TRIAL: NCT05062044
Title: Prospective International Multicenter Observational Cohort Study Evaluating Progress and Outcomes of Pregnancy in Women Using Various Vitamin Support Regimens Before and During Pregnancy (UNONA Study)
Brief Title: A Study to Gather Information About the Progress and Outcomes of Pregnancy in Women Using Various Vitamin Support Plans Before and During Pregnancy
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21967
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Prevention of Vitamin Deficiency During and/or Before Pregnancy
Keywords: Preconceptional preparation; Pregnancy; Folic acid; Multivitamins; Vitamin deficiency; Supplementation; Anemia during pregnancy; Fetus growth and development
MeSH Terms: conditions — Avitaminosis | interventions — Geritol; Folic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Multivitamins usage in pregravidal preparation: Participants start use of Elevit multiple micronutrient (MMN) before pregnancy.
  Interventions: Dietary Supplement: Multivitamins (Elevit, BAY987808); Dietary Supplement: Multivitamins (Elevit, BAY2906300); Drug: Multivitamins (Elevit, BAY987386)
- Multivitamins usage during pregnancy: Participants start use of Elevit multiple micronutrient (MMN) in the first trimester of pregnancy.
  Interventions: Dietary Supplement: Multivitamins (Elevit, BAY987808); Dietary Supplement: Multivitamins (Elevit, BAY2906300); Drug: Multivitamins (Elevit, BAY987386)
- Folic acid usage during pregnancy: Participants use folic acid in accordance with clinical guidelines.
  Interventions: Dietary Supplement: Folic acid

INTERVENTIONS:
Dietary Supplement: Multivitamins (Elevit, BAY987808) — Following the manner of observational study, no intervention will be provided in the study. Participants follows approved clinical guidelines, without interference by the study initiator or study protocol.
  Other Names: Elevit® planning and the first trimester
  Groups: Multivitamins usage during pregnancy; Multivitamins usage in pregravidal preparation
Dietary Supplement: Multivitamins (Elevit, BAY2906300) — Following the manner of observational study, no intervention will be provided in the study. Participants follows approved clinical guidelines, without interference by the study initiator or study protocol.
  Other Names: Second and Third Trimesters under Elevit®
  Groups: Multivitamins usage during pregnancy; Multivitamins usage in pregravidal preparation
Drug: Multivitamins (Elevit, BAY987386) — Following the manner of observational study, no intervention will be provided in the study. Participants follows approved clinical guidelines, without interference by the study initiator or study protocol.
  Other Names: Elevit® Pronatal
  Groups: Multivitamins usage during pregnancy; Multivitamins usage in pregravidal preparation
Dietary Supplement: Folic acid — Following the manner of observational study, no intervention will be provided in the study. Participants follows approved clinical guidelines, without interference by the study initiator or study protocol.
  Groups: Folic acid usage during pregnancy

SUMMARY:
This is an observational study in which data from the participants who will be taking different vitamin supplementation regimes before and during pregnancy.

Vitamin deficiency is a condition where there is not enough vitamins in the body. During pregnancy, a woman's body may require more vitamins than usual. When the body does not get enough vitamins, people can take vitamin supplements to help increase the amount of vitamins in the body.

It is already known, that polyvitamins can decrease risks of anemia (low level of red cells in the blood), neural tube defects (severe congenital anomaly of neural system) or other malformations, but also on several pregnancy complications.

Nevertheless, a significant amount of evidence on the use of vitamins during pregnancy has been obtained in countries with low and middle level of living standards.

Countries with higher living standards may have different prevalence of vitamin insufficiency, thereby it is not clearly known how vitamin supplementation may help to reduce pregnancy complications in these population. So, researchers think it is important to do more studies.

Elevit contains many different vitamins and minerals. These vitamins and minerals are important to help women before and during pregnancy.

In this study, the researchers want to collect more data about how well pregnancies progress and the outcomes of the pregnancies in women who are taking different vitamin treatment or supplements, including elevit.

To do this, the researchers will review information collected from the participants to:

* calculate how many women give birth without any complications between weeks 37 and 42 of their pregnancies
* calculate how many women have low levels of red blood cells in the blood during the third trimester of their pregnancies
* calculate how many women have a serious condition called preeclampsia during their pregnancy, a condition in which pregnant women have a sudden rise in blood pressure and swelling in the hands, feet and face
* calculate how many women give birth to babies who weigh less than expected at the time of their birth
* give the women a questionnaire to complete during each trimester to see how they are feeling

The participants will have decided with their doctor to start their vitamin treatment or supplements before getting pregnant or during their pregnancy.

During the study, the researchers will collect the women's information from their medical records taken during their regular medical appointments. The study will include women who are pregnant and who are planning to get pregnant. The study will include both women who have vitamin deficiency and women who do not have vitamin deficiency.

Each participant will be in this study for up to 18 months., The whole study will last about 2 years and 10 months. During this time, the participants will visit their doctor 5 times as part of their usual care. The study is planned to collect data from October 2021 until June 2024.

ELIGIBILITY:
Inclusion Criteria:

* A woman aged 18 through 45 (inclusive) who is planning a pregnancy or with an already confirmed pregnancy with pregnancy term up to 12 weeks (pregnancy was confirmed by laboratory and/or ultrasound method).
* Decision to use Elevit® MMN or monocomponent supplementation of folic acid was made independent of study participation, and made prior to inclusion into this study.
* Provided signed Informed Consent to participate in the study
* Ability to understand and follow study-related instructions.
* Be willing and able to participate in all scheduled visits, treatment plan, laboratory tests and other trial procedures according to the study protocol and the standard medical practice.

Exclusion Criteria:

* Concurrent participation in interventional or other non-interventional study.
* The gestation period is more than 12 weeks.
* Taking any folate-containing products other than Elevit® for three months prior to enrollment in the study.
* Usage of other than Elevit Multiple Micronutrient product.
* Malignant neoplasms at present or in history.
* History of pregnancy with congenital malformations.
* Contraindications to the use of MMN Elevit specified in the approved instructions for use (for the medicinal product "Elevit® Pronatal") or leaflet (for dietary supplements "Elevit® planning and first trimester" and dietary supplements "Second and Third Trimester" of the trademark " Elevit®").
* Concomitant diseases in the stage of decompensation.
* Multiple pregnancy diagnosed before enrollment.
* Other pathological conditions that make it impossible for the subject to participate in the program (by the decision of the attending physician).
* Member or first-degree relative of study staff or the Sponsor directly involved in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women aged 18 through 45 (inclusive) planning a pregnancy or with an already confirmed pregnancy (pregnancy was confirmed using laboratory and/or instrumental methods, pregnancy term is up to 12 weeks), of different risk of having micronutrient insufficiency and using Elevit Multiple Micronutrient (MMN) or a monocomponent supplementation with folic acid and being in compliance with the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-04-13 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with normally completed pregnancies | Up to 18 months
  Normally completed pregnancy is defined as pregnancies completed in term 37-42 weeks inclusive, with no major pregnancy maternal and fetus complications such as severe maternal anemia, preeclampsia, congenital anomalies, fetal growth retardation or other pregnancy complication concerned by the study investigator.
Number of participants with maternal anemia of any severity in third trimester (hemoglobin [Hb] <110 g/L) | Up to 18 months
Number of participants with preeclampsia of any severity | Up to 18 months
  Preeclampsia is defined (arterial hypertension blood pressure [BP]>= 140/90 mmHg) in combination with proteinuria (≥0.3 g/l in daily urine) after the 20th week of pregnancy); OR in absence of proteinuria with new onset of the following: Signs of multiple organ failure; Thrombocytopenia: platelet count less than 100,000 x 10^9 /L; Serum creatinine > 1.1 mg/dL or doubling of the serum creatinine; Elevated liver transaminases to twice normal; Pulmonary edema; New onset headache unresponsive to medication; Visual symptoms.
Number of participants with small-for-gestational newborns | Up to 18 months
  Small for gestational age is defined as a newborn with weigh less than 10th percentile of normal weigh for gestational age.
Number of participants having low and very low birth weight newborns | Up to 18 months
  Low birth weight is a term used to describe babies who are born weighing less than 5 pounds, 8 ounces (2,500 grams). Babies weighing less than 3 pounds, 5 ounces (1,500 grams) at birth are considered as very low birth weight.
Mean and change in score of quality of life gravidarum (QoL-Grav) in first to third trimester | Up to 12 months
  QoL-Grav questionnaire is designed for assessing the quality of life during pregravidal preparation and during pregnancy. The overall score normally varies from 15 to 35, the lower the score, the higher the quality of life.

SECONDARY OUTCOMES:
Number and severity of anemia at any trimesters | Up to 18 months
Number of usage of iron medications for the purposes of anemia | Up to 12 months
Change of anemia severity from first to third trimester | Up to 12 months
Number of participants with preterm birth | Up to 12 months
  Preterm birth is defined as a childbirth that occurred at a period of 22 to 37 complete weeks and with a fetal weight of more than 500g.
  Extremely preterm birth: 28 complete weeks; Early preterm birth: 28 to 32 weeks; Moderate to late preterm: 32 to 37 weeks.
Number of participants with fetal growth restriction during third trimester | Up to 12 months
  Fetal growth restriction (FGR) is a condition in which an unborn baby (fetus) is smaller than expected for the number of weeks of pregnancy (gestational age). It is described as an estimated weight less than the 10th percentile. FGR will be assessed by ultrasonography specialist during usual ultrasound examination in 3rd trimester.
Number of participants with post-term birth | Up to 12 months
  Post-term pregnancy is defined as pregnancy that has extended to or beyond 42 weeks of gestation (294 days).
Number of participants with gestational diabetes | Up to 12 months
Number of participants with confirmed glucose intolerance during third trimester | Up to 12 months
Number of participants with congenital malformations | Up to 12 months
  Congenital malformations will be defined as any anomalies in the development of the fetus, classified as malformations and coded in ICD-10 as "Congenital anomalies [malformations], deformities and chromosomal disorders (Q00-Q99)".
Number of participants with fetal macrosomia | Up to 12 months
  Large fetus defined as birth weight > 4000 g, provided that it is not caused by various congenital neoplasms and other fetal diseases (erythroblastosis, teratoma, hydrocephalus, etc.).
Number of participants with excessive vomiting in pregnant women | Up to 12 months
  Vomiting occur in every third pregnancy, in 90% cases it is normal course of pregnancy and happens no more than 2-3 times a day, more often on an empty stomach, and does not violate the general condition of pregnant woman.
Number of pregnancy within 6 months of periconceptional supplementation in women with different levels of fertile function | Up to 18 months
  In age groups up to 35 years and 35 years and older, with the presence of concomitant gynecological pathology (menstrual irregularities, inflammatory processes in the pelvic area, anomalies in development of genital organs, history of uterine surgery, endometriosis, obesity, hyper- and hypothyroidism, autoimmune diseases)
Number of participants with spontaneous abortion/miscarriage | Up to 12 months
  Spontaneous miscarriage is the loss of pregnancy naturally before twenty weeks of gestation.
Normal weight gain in newborns in the first month of life in accordance with WHO child growth standards | Up to 12 months
  WHO stands for world health organization.
Number of participants with exclusive breastfeeding, mixed and artificial feeding in the first month after delivery | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gennady T. Sukhikh, Dr. Medical Science, Professor, Study Chair — Federal State Budgetary Institution "National Medical Research Center for Obstetrics, Gynecology and Perinatology named after Academician V.I. Kulakov" Ministry of Health of the Russian Federation.
Locations (3):
- Many Locations, Multiple Locations, Kazakhstan
- Many Locations, Multiple Locations, Russia
- Many Locations, Multiple Locations, Uzbekistan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.